CLINICAL TRIAL: NCT00282724
Title: A Randomized, Double-blind, Placebo-controlled Phase II/III Trial to Evaluate the Efficacy and Safety of 2 Doses of Oral Liarozole (75 mg od and 150 mg od) Given During 12 Weeks in Lamellar Ichthyosis
Brief Title: Efficacy and Safety of Two Doses of Liarozole vs. Placebo for the Treatment of Lamellar Ichthyosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BT0500INT001
Record Dates: First submitted 2006-01-20; First posted 2006-01-27 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Ichthyosis, Lamellar
Keywords: Lamellar ichthyosis; Liarozole; Investigator's Global Assessment; Scaling
MeSH Terms: conditions — Ichthyosis, Lamellar | interventions — liarozole

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Liarozole

SUMMARY:
Lamellar ichthyosis is a congenital disease of the skin with a generalized scaling. The primary activity of liarozole is considered to be the inhibition of the degradation of a substance called retinoic acid, which is the principal endogenous regulator of growth and differentiation of epithelial tissues in mammals. The current study intends to evaluate the efficacy and safety in patients with lamellar ichthyosis.

DETAILED DESCRIPTION:
Lamellar ichthyosis is an autosomal recessive disorder that is apparent at birth and is present throughout life. Although the disorder is not life threatening, it is quite disfiguring and causes considerable psychological stress to affected patients. Prevalence is less than 1 case per 300,000 individuals. Treatment is mainly symptomatic i.e. emollients with or without keratolytic agents. Treatment with systemic retinoids is reserved for those patients, refractory to conventional therapy, because of the long-term adverse effects and teratogenicity of systemic retinoids.

Liarozole may provide a new concept for the treatment of this condition. Because of its mechanism of action, retinoic acid (RA) levels will only be increased in tissues that are targets for RA production.

The proposed Phase II/III study intends to evaluate the efficacy of liarozole compared with placebo, in patients with lamellar ichthyosis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either sex aged 14 years or older.
* Clinical diagnosis of lamellar ichthyosis
* Women of childbearing potential should use appropriate contraception
* Women of childbearing potential should have a negative pregnancy test at screening visit.
* Subjects are, except for their lamellar ichthyosis, in good general health.
* Subjects and legal representative(s), if applicable, signed informed consent.

Exclusion Criteria:

* Subject is receiving topical (except emollient), UV treatment or systemic treatment for ichthyosis.
* Subject is pregnant or breast feeding.
* History or suspicion of alcohol or drug abuse.
* Significant co-existing diseases.
* Clinically significant abnormal ECG
* History of hypersensitivity to retinoids or any of the ingredients in the trial medication.
* Clinically relevant laboratory abnormalities at screening.
* Use of immune-suppressive drugs including topical or systemic corticosteroids.
* Participation in an investigational trial 30 days prior to the start of the trial.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2006-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Efficacy: Investigator's Global Assessment

SECONDARY OUTCOMES:
Overall Scaling Score
Severity scores of other symptoms
Quality of Life
Safety and tolerability
Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Koen van Rossem, MD, PhD, Study Director — Barrier Therapeutics/ Stiefel, a GSK Company
Locations (16):
- Belgium (2):
  - Academisch Ziekenhuis Vrije Universiteit Brussel, Brussels
  - Geel, Geel
- Canada (2):
  - Hôpital Saint-Justine, Montreal
  - Newlab Clinical Research Inc., St. John's
- Instituto Dermatologico, Santo Domingo, Dominican Republic
- Hôtel Dieu CHU, Nantes, France
- Germany (4):
  - Tomesa Fachklinik, Bad Salzschlirf
  - Dueren, Düren
  - Otto-von-Guericke-Universität, Magdeburg
  - University Hospital Muenster, Münster
- Italy (2):
  - Fondazione Policlinico Mangiagalli e Regina Elena, Milan
  - Istituto Dermopatico dell'Immacolata, Rome
- Netherlands (2):
  - Academisch Ziekenhuis Maastricht, Maastricht
  - University Hospital Rotterdam, Rotterdam
- Rikshospitalet Universitetsklinikk, Oslo, Norway
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Background] Van Wauwe JP, Coene MC, Goossens J, Cools W, Monbaliu J. Effects of cytochrome P-450 inhibitors on the in vivo metabolism of all-trans-retinoic acid in rats. J Pharmacol Exp Ther. 1990 Jan;252(1):365-9. PMID 2299598
- [Background] Van Wauwe J, Van Nyen G, Coene MC, Stoppie P, Cools W, Goossens J, Borghgraef P, Janssen PA. Liarozole, an inhibitor of retinoic acid metabolism, exerts retinoid-mimetic effects in vivo. J Pharmacol Exp Ther. 1992 May;261(2):773-9. PMID 1374473
- [Background] Van Wauwe J, Coene MC, Cools W, Goossens J, Lauwers W, Le Jeune L, Van Hove C, Van Nyen G. Liarozole fumarate inhibits the metabolism of 4-keto-all-trans-retinoic acid. Biochem Pharmacol. 1994 Feb 11;47(4):737-41. doi: 10.1016/0006-2952(94)90137-6. PMID 8129749
- [Background] Kang S, Duell EA, Kim KJ, Voorhees JJ. Liarozole inhibits human epidermal retinoic acid 4-hydroxylase activity and differentially augments human skin responses to retinoic acid and retinol in vivo. J Invest Dermatol. 1996 Aug;107(2):183-7. doi: 10.1111/1523-1747.ep12329579. PMID 8757760
- [Background] Dockx P, Decree J, Degreef H. Inhibition of the metabolism of endogenous retinoic acid as treatment for severe psoriasis: an open study with oral liarozole. Br J Dermatol. 1995 Sep;133(3):426-32. doi: 10.1111/j.1365-2133.1995.tb02672.x. PMID 8546999
- [Background] Berth-Jones J, Todd G, Hutchinson PE, Thestrup-Pedersen K, Vanhoutte FP. Treatment of psoriasis with oral liarozole: a dose-ranging study. Br J Dermatol. 2000 Dec;143(6):1170-6. doi: 10.1046/j.1365-2133.2000.03884.x. PMID 11122017
- [Background] Bhushan M, Burden AD, McElhone K, James R, Vanhoutte FP, Griffiths CE. Oral liarozole in the treatment of palmoplantar pustular psoriasis: a randomized, double-blind, placebo-controlled study. Br J Dermatol. 2001 Oct;145(4):546-53. doi: 10.1046/j.1365-2133.2001.04411.x. PMID 11703279
- [Background] Lucker GP, Heremans AM, Boegheim PJ, van de Kerkhof PC, Steijlen PM. Oral treatment of ichthyosis by the cytochrome P-450 inhibitor liarozole. Br J Dermatol. 1997 Jan;136(1):71-5. PMID 9039298
- [Derived] Vahlquist A, Blockhuys S, Steijlen P, van Rossem K, Didona B, Blanco D, Traupe H. Oral liarozole in the treatment of patients with moderate/severe lamellar ichthyosis: results of a randomized, double-blind, multinational, placebo-controlled phase II/III trial. Br J Dermatol. 2014 Jan;170(1):173-81. doi: 10.1111/bjd.12626. PMID 24102348